CLINICAL TRIAL: NCT05011851
Title: An Open-Label Study of the Safety, Tolerability, and Pharmacokinetics of Oral NNZ-2591 in Angelman Syndrome
Acronym: AS-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuren Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU-2591-AS-001
Record Dates: First submitted 2021-08-05; First posted 2021-08-18 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Angelman Syndrome
Keywords: Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome | interventions — cyclo-L-glycyl-L-2-allylproline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NNZ-2591 (Experimental): NNZ-2591 oral solution (50mg/mL) to be administered twice daily for 13 weeks.
  Interventions: Drug: NNZ-2591

INTERVENTIONS:
Drug: NNZ-2591 — NNZ-2591 oral solution (50mg/mL) to be administered twice daily for 13 weeks.
  Other Names: Cyclo-L-Glycyl-L-2-Allylproline

SUMMARY:
A study of the safety, tolerability and pharmacokinetics of NNZ-2591 and measures of efficacy in children and adolescents with Angelman syndrome

DETAILED DESCRIPTION:
The primary purpose of this study is to investigate the safety, tolerability and pharmacokinetics of treatment with NNZ-2591 oral solution, 50mg/L, in children and adolescents with Angelman syndrome. The secondary purpose is to investigate measures of efficacy of subjects will receive treatment of 50mg/mL orally administered NNZ-2591 for a total of 13 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of AS with a documented disease-causing genetic etiology known to impact maternally derived UBE3A expression in brain.
2. Males or females aged 3-17 years
3. Body Weight of >12Kg
4. Subjects with a Clinical Global Impression - Severity (CGI-S) score of 3 or greater
5. Not actively undergoing regression or loss of skills, defined as no persistent loss of previously acquired developmental skills for a period within 3 months of the Screening visit
6. Each subject must be able to swallow the study medication provided as a liquid solution.
7. Caregiver(s) must have sufficient English language skills.

Exclusion Criteria:

1. Mosaicism for disease-causing mutation.
2. Clinically Significant abnormalities in safety laboratory testing or vital signs at screening
3. Abnormal QTcF interval or prolongation at Screening.
4. Positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and previous COVID 19 infection with last 12 months that required hospitalization.
5. Unstable or changes to Psychotropic treatment 2 weeks prior to screening .
6. Excluded concomitant treatments
7. Actively undergoing regression or loss of skills.
8. Unstable seizure profile.
9. Current clinically significant renal conditions and abnormalities
10. Current clinically significant cardiovascular, hepatic, gastrointestinal, respiratory, endocrine disease, or clinically significant organ impairment.
11. Current clinically significant hypo or hyperthyroidism, Type 1 or Type 2 diabetes mellitus requiring insulin (whether well controlled or uncontrolled), or uncontrolled Type 1 or Type 2 diabetes.
12. Has planned surgery during the study.
13. History of, or current, cerebrovascular disease or brain trauma.
14. History of, or current catatonia or catatonia-like symptoms.
15. History of, or current, malignancy.
16. Current major or persistent depressive disorder (including bipolar depression).
17. Significant, uncorrected visual or uncorrected hearing impairment.
18. Allergy to strawberry.
19. Positive pregnancy test
20. Subject is judged by the Investigator or Medical Monitor to be inappropriate for the study

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 13 weeks
  To examine the incidence, severity and frequency of adverse events (AEs), including serious adverse events (SAEs) during treatment with NNZ-2591.
Pharmacokinetic - Typical AUC24 of 30kg Child | 13 weeks
  Area under the concentration-time curve of NNZ-2591 over 24 hours
Pharmacokinetic - Typical t1/2 in 30 kg Child | 13 weeks
  Apparent terminal elimination half-life of NNZ-2591

SECONDARY OUTCOMES:
Angelman syndrome-specific Clinical Global Impression Scale-Overall Improvement (CGI-I) | 13 weeks
  Assessed by Angelman syndrome-specific Clinical Global Impression Scale-Overall Improvement (CGI-I). Score on a Likert scale (1-7) where lower scores are better
Caregiver Impression of Improvement : Overall Score | 13 weeks
  Caregiver Impression of Improvement: Overall Score. Measured on a 7-point Likert scale (1-7) where lower scores are better.
Angelman syndrome-specific Clinical Global Impression Scale - Severity (CGI-S): Overall Score | 13 weeks
  Angelman syndrome-specific Clinical Global Impression Scale-Severity (CGI-S): Change from baseline on overall score based on a 7-point Likert scale (1-7) where lower scores are better.
Angelman syndrome Clinician Domain Specific Rating Scale (AS-DSRS) | 13 weeks
  Angelman syndrome Clinician Domain Specific Rating Scale (AS-DSRS). Change from baseline in total score based on a 5-point Likert scale (0-4) where lower scores are better.
Caregiver Top 3 Concerns | 13 weeks
  Caregiver Top 3 Concerns: Change from baseline in Average Concerns Severity.
MacArthur-Bates Communicative Development Inventory (MB-CDI) | 13 weeks
  MacArthur-Bates Communicative Development Inventory (MB-CDI)
Observer-Reported Communication Ability (ORCA) | 13 weeks
  Observer-Reported Communication Ability (ORCA). Change from baseline in modified t-score. Scores range from 25.8 - 83.8 with higher scores indicating greater communication abililty. A positive change from baseline indicates improvement
Aberrant Behavior Checklist-2 (ABC-2) | 13 weeks
  Aberrant Behavior Checklist-2 (ABC-2) - Change from baseline in total score. Higher scores indicate more behavioral issues. A negative change from baseline indicates improvement.
Child Sleep Habits Questionnaire (CSHQ) | 13 weeks
  Child Sleep Habits Questionnaire (CSHQ). Change from baseline in total score. Range of scores was (33-99) with higher scores being worse
Gastrointestinal Health Questionnaire (GIHQ) | 13 weeks
  Gastrointestinal Health Questionnaire (GIHQ)
Vineland Adaptive Behavior Scales-3, Interview version | 13 weeks
  Vineland Adaptive Behavior Scales-3, Interview version; Composite standard score
Exploratory efficacy measurement | 13 weeks
  Assessed by Bayley Scales of Infant Development-4, Vineland Motor subscales
Quality of Life Inventory-Disability (QI-Disability) | 13 weeks
  Quality of Life Inventory-Disability (QI-Disability). Change from baseline inoverall score. Scores range from 0-100 with higher scores indicating better quality of life. A positive change indicates improvement
Impact of Childhood Neurological Disability (ICND) | 13 weeks
  Impact of Childhood Neurological Disability (ICND): Change from baseline in overall quality of life rating. Scores range from 1-6, with a higher score indicating better quality of life. A positive change from baseline indicates improvement

CONTACTS AND LOCATIONS:
Overall Officials: James Shaw, Study Director — Neuren Pharmaceuticals
Locations (3):
- Australia (3):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Centre for Clinical Trials in Rare Neurodevelopmental Disorders at Children's Health Queensland Hospital and Health Service, South Brisbane, Queensland
  - Austin Health, Heidelberg, Victoria

IPD SHARING:
Plan to Share IPD: No